CLINICAL TRIAL: NCT00272922
Title: Randomized, Prospective Controlled Trial of Paraesophageal Hernia Repair With Small Intestinal Submucosa (SIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-1931-A-01 (Institution #)
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Hernia; Paraesophageal Hernia
Keywords: Biomaterials; Paraesophageal Hernia; Laparoscopy
MeSH Terms: conditions — Hernia; Hernia, Hiatal | interventions — Herniorrhaphy

INTERVENTIONS:
Device: hernia repair

SUMMARY:
The purpose of this randomized study is to determine whether a type of mesh derived from a layer of pig small intestine (SIS) is of benefit in treating paraesophageal hernias versus standard surgical suture repair.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Documented symptomatic paraesophageal hernia
* Ability to participate in follow-up evaluation
* Has a telephone
* Free of cognitive or speech impairment

Exclusion Criteria:

* Patients requiring intra-operative conversion to an open procedure
* Unable to close the crura primarily
* Short esophagus that requires the surgeon to perform a lengthening procedure
* Previous operation of the esphagus or stomach
* Associated gastrointestinal diseases that require extensive medical or surgical intervention that might interfere with quality of like assessment
* Intraoperative full-thickness perforation of the esophagus
* Emergent operation for acute volvulus
* Ineffective peristalsis defined as average amplitude of peristalsis less than 30 mmHg or < 70% propagation of peristaltic waves in the distal esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant K Oelschlager, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States